CLINICAL TRIAL: NCT02909322
Title: Analgesic and Hemodynamic Effects of Continuous Epidural Analgesia Compared to Paravertebral Block in Liver Resection Patients
Brief Title: Epidural Versus Paravertebral Block Analgesia After Hepatectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Anthony Ho (Other)
Responsible Party: Sponsor-Investigator, Dr. Anthony Ho, Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANAE-270-15
Record Dates: First submitted 2016-07-13; First posted 2016-09-21 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Pain Control After Elective Hepatectomy
MeSH Terms: interventions — Bupivacaine; Hydromorphone; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Epidural Analgesia (Active Comparator): Analgesic medications will be given via epidural, the standard of care.
  Interventions: Procedure: Bupivacaine and Hydromorphone
- Paravertebral Block Analgesia (Experimental): Analgesic medications will be given via the paravertebral space.
  Interventions: Procedure: Ropivacaine and Hydromorphone

INTERVENTIONS:
Procedure: Bupivacaine and Hydromorphone — Patients receive bupivacaine and hydromorphone infusion and bolus doses during surgery and 3 days after surgery.
  Arms: Continuous Epidural Analgesia
Procedure: Ropivacaine and Hydromorphone — Patients receive ropivacaine and hydromorphone infusion and bolus doses during surgery and 3 days after surgery.
  Arms: Paravertebral Block Analgesia

SUMMARY:
The best mode of analgesia delivery after hepatectomy is currently unknown. Many institutions routinely use continuous epidural analgesia (CEA) for pain control in this patient population. A functioning CEA provides adequate analgesia, but is associated with high failure rates (20-30%) and sometimes significant hemodynamic disturbances (hypotension) requiring an increased amount of intravenous fluid and blood products to maintain homeostasis. Furthermore, its safety has been the subject of debate in liver resection patients due to the elevated risk of epidural hematoma and its serious neurological consequences. These limitations highlight the need to explore other options for analgesic control after hepatectomy, such as paravertebral block (PVB). PVB has been shown to provide similar analgesia with a lower incidence of pulmonary complications, side effects (pruritis, urinary retention, nausea and vomiting, hypotension), and failure rates (6.1%) when compared to CEA in thoracic surgery, and therefore has been suggested as a safer alternative in hepatectomy patients. Despite this, there are no studies comparing the efficacy of CEA and PVB as analgesic techniques after hepatectomy. The investigators propose a randomized controlled trial to compare the analgesic efficacy, side effects, and complications associated with CEA and PVB in patients undergoing elective hepatectomy through a right subcostal incision.

DETAILED DESCRIPTION:
The best mode of analgesia delivery after hepatectomy is currently unknown. Many institutions routinely use continuous epidural analgesia (CEA) for pain control in hepatectomy patients. However, its safety has been the subject of debate. Paravertebral block (PVB) has been suggested as a safer alternative in this patient population. Despite this, there are no studies comparing the efficacy of CEA and PVB as analgesic techniques after hepatectomy. Although CEA provides high quality analgesia, and reduces cardiovascular and respiratory complications and the incidence of postoperative thromboembolic events, it is associated with hypotension and complications such as epidural hematoma, epidural abscess, and spinal cord injury, which are serious concerns in hepatectomy patients. Furthermore, patients given CEA are more likely to need blood transfusions, and transfused patients have significantly higher mortality rates, complications related to infection, and hospital length of stay. PVB is a less popular technique that involves injecting local anesthetic (LA) into the paravertebral space. This technique has been successfully used for pain relief after several surgical procedures, including ablation of hepatic tumours and hepatectomy. Although CEA and PVB have never been compared in hepatectomy patients, they have been compared in thoracotomy patients; in this patient population, PVB and CEA provide similar levels of pain control, but CEA is associated with more complications and side effects such as hypotension, nausea, vomiting, and urinary retention, and PVB is associated with better pulmonary function. Both CEA and PVB are reasonably effective for post-hepatectomy analgesia compared to placebo, and have their own strengths and weaknesses. The gold standard CEA provides excellent analgesia at the expense of more intense hypotension, significant failure rates (20-30%), and a higher risk of epidural hematoma and its serious neurological consequences. These limitations highlight the need to explore other options for analgesic control after hepatectomy such as PVB. Therefore, the investigators propose a randomized controlled trial to compare the analgesic efficacy, hemodynamic changes, and side effects in CEA and PVB in patients undergoing elective hepatectomy through a right subcostal incision. Since CEA is currently the gold standard for analgesia after hepatectomy, the investigators propose a non-inferiority trial to determine whether PVB produces a similar analgesic profile to CEA in hepatectomy patients, while being associated with fewer adverse side effects.

This is a randomized, controlled, pilot study. It will consist of two groups of participants undergoing hepatectomy: those receiving CEA, and those receiving PVB for analgesic control. CEA and PVB protocols will follow the usual standard of care at Kingston General Hospital (KGH). Participants in the CEA group will receive bupivacaine with hydromorphone infusion after induction of general anesthesia for surgery. Participants in the PVB group will receive a bolus dose of ropivacaine, and then ropivacaine infusion after induction of general anesthesia. Upon emergence from anesthesia, all participants will be transferred to the post-anesthetic care unit (PACU). Here, CEA participants will be started on patient-controlled epidural analgesia (PCEA) of bupivacaine and hydromorphone plus a self-administered bolus dose with a lockout period of 30 min if participants require additional pain relief, and PVB participants will be started on a patient-controlled paravertebral analgesia (PCPA) of ropivacaine plus a self-administered bolus dose with a lockout period of 30 min if participants require additional pain relief. All participants will receive oral hydromorphone every 4 hours as required for breakthrough pain relief starting on the morning of the second postoperative day. A member of the research team will assess the presence and severity of pain and nausea during the postoperative period. The assessments will be performed at 30 minutes after arrival to the PACU, and thereafter at 4, 8, 24, 48, and 72 hours after surgery. Investigators will ask all participants to score their pain at rest and with coughing on a numeric rating scale (NRS, where 0=no pain and 10=worst pain imaginable), and nausea scores (0=none, 1=mild, 2=moderate, 3=vomiting) at each of the above listed time points. At 72 hours after surgery, participant satisfaction with regard to analgesia will be assessed (1=very poor, 2=poor, 3=satisfactory, 4=good, 5=excellent). The requirement for breakthrough pain relief, the time of first breakthrough pain relief request, and cumulative opioid consumption will be recorded during the postoperative 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* ASA I-III
* Undergoing elective liver resection through right subcostal incision
* Proficient in English
* Competent to give consent

Exclusion Criteria:

* Not given informed consent
* Not competent to give informed consent
* Dementia or neurological impairment
* Jaundice (bilirubin > 50μmol/L)
* Liver resection combined with secondary surgical procedure
* Contraindication to either epidural or paravertebral block (INR ≥ 1.6, platelet count < 100,000/mm3, fever, previous back surgery)
* Anticipated significant coagulopathy post-liver resection (as indicated by a Model for End-Stage Liver Disease score >8 or predicted liver resection of more than 500g)
* Contraindications to any of the study medications
* Remain intubated in the postoperative period, due to inability to assess pain scores
* Midline incision and/or any type of extended incision that is not restricted to the standard right subcostal incision
* Body mass index < 18 or > 40
* Pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 0-72 hours after surgery
  Cumulative opioid consumption during the postoperative period will be recorded.
Time to first request for opioids | 0-72 hours after surgery
  The first time after surgery each participant asks for opioid medication for pain will be recorded.
Pain scores | 30min, 4, 8, 24, 48, and 72 hours after surgery
  At the specified time points, participants will rate their pain on a scale from 0 to 10.

SECONDARY OUTCOMES:
Nausea | 30min, 4, 8, 24, 48, and 72 hours after surgery
  At the specified time points, participants will rate their nausea.
Satisfaction with analgesia | 72 hours after surgery
  Participants will rate their satisfaction with their analgesia.
Success rates of CEA and PVB | 0-72 hours after surgery
  The number of successful CEA and PVB procedures will be recorded.
Failure rates of CEA and PVB | 0-72 hours after surgery
  The number of therapeutic failures of CEA and PVB procedures will be recorded.
Mean arterial pressure | 0-72 hours after surgery
  Mean arterial pressure will be recorded.
Central venous pressure | 0-72 hours after surgery
  Central venous pressure will be recorded.
Urine output | 0-72 hours after surgery
  Urine output will be recorded.
Acid-base | 0-72 hours after surgery
  pH, bicarbonate, partial pressure of carbon dioxide, and partial pressure of oxygen in the blood will be recorded.
Intravenous fluid volume | 0-72 hours after surgery
  Total volume of crystalloids, colloids, and blood products given perioperatively and during the 72 hours after surgery will be recorded.
Vasopressor volume | 0-72 hours after surgery
  Total volume of vasopressors given perioperatively and during the 72 hours after surgery will be recorded.
Resumption of full oral diet | 0-72 hours after surgery
  The number of days taken to resume a full oral diet will be recorded.
Hospital length of stay | 0-72 hours after surgery
  The number of days until participants are discharged will be recorded.
Adverse events | 0-72 hours after surgery
  Any postoperative adverse events will be recorded.
Demographic data | Upon enrollment up to 72 hours after surgery
  Descriptive demographic data will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony MH Ho, MD,FRCPC, Principal Investigator — Queen's University/ Kingston Health Sciences Centre
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Page A, Rostad B, Staley CA, Levy JH, Park J, Goodman M, Sarmiento JM, Galloway J, Delman KA, Kooby DA. Epidural analgesia in hepatic resection. J Am Coll Surg. 2008 Jun;206(6):1184-92. doi: 10.1016/j.jamcollsurg.2007.12.041. Epub 2008 Apr 14. PMID 18501817
- [Background] Siniscalchi A, Begliomini B, De Pietri L, Braglia V, Gazzi M, Masetti M, Di Benedetto F, Pinna AD, Miller CM, Pasetto A. Increased prothrombin time and platelet counts in living donor right hepatectomy: implications for epidural anesthesia. Liver Transpl. 2004 Sep;10(9):1144-9. doi: 10.1002/lt.20235. PMID 15350005
- [Background] Choi SJ, Gwak MS, Ko JS, Kim GS, Ahn HJ, Yang M, Hahm TS, Lee SM, Kim MH, Joh JW. The changes in coagulation profile and epidural catheter safety for living liver donors: a report on 6 years of our experience. Liver Transpl. 2007 Jan;13(1):62-70. doi: 10.1002/lt.20933. PMID 17192873
- [Background] Matot I, Scheinin O, Eid A, Jurim O. Epidural anesthesia and analgesia in liver resection. Anesth Analg. 2002 Nov;95(5):1179-81, table of contents. doi: 10.1097/00000539-200211000-00009. PMID 12401587
- [Background] Shontz R, Karuparthy V, Temple R, Brennan TJ. Prevalence and risk factors predisposing to coagulopathy in patients receiving epidural analgesia for hepatic surgery. Reg Anesth Pain Med. 2009 Jul-Aug;34(4):308-11. doi: 10.1097/AAP.0b013e3181ac7d00. PMID 19574863
- [Background] Kehlet H, Holte K. Effect of postoperative analgesia on surgical outcome. Br J Anaesth. 2001 Jul;87(1):62-72. doi: 10.1093/bja/87.1.62. No abstract available. PMID 11460814
- [Background] Stamenkovic DM, Jankovic ZB, Toogood GJ, Lodge JP, Bellamy MC. Epidural analgesia and liver resection: postoperative coagulation disorders and epidural catheter removal. Minerva Anestesiol. 2011 Jul;77(7):671-9. Epub 2008 Nov 27. PMID 19037193
- [Background] Cook TM, Counsell D, Wildsmith JA; Royal College of Anaesthetists Third National Audit Project. Major complications of central neuraxial block: report on the Third National Audit Project of the Royal College of Anaesthetists. Br J Anaesth. 2009 Feb;102(2):179-90. doi: 10.1093/bja/aen360. Epub 2009 Jan 12. PMID 19139027
- [Background] Weinberg L, Scurrah N, Gunning K, McNicol L. Postoperative changes in prothrombin time following hepatic resection: implications for perioperative analgesia. Anaesth Intensive Care. 2006 Aug;34(4):438-43. doi: 10.1177/0310057X0603400405. PMID 16913338
- [Background] Wong-Lun-Hing EM, van Dam RM, Welsh FK, Wells JK, John TG, Cresswell AB, Dejong CH, Rees M. Postoperative pain control using continuous i.m. bupivacaine infusion plus patient-controlled analgesia compared with epidural analgesia after major hepatectomy. HPB (Oxford). 2014 Jul;16(7):601-9. doi: 10.1111/hpb.12183. Epub 2013 Oct 23. PMID 24151899
- [Background] Revie EJ, Massie LJ, McNally SJ, McKeown DW, Garden OJ, Wigmore SJ. Effectiveness of epidural analgesia following open liver resection. HPB (Oxford). 2011 Mar;13(3):206-11. doi: 10.1111/j.1477-2574.2010.00274.x. PMID 21309939
- [Background] McLeod G, Davies H, Munnoch N, Bannister J, MacRae W. Postoperative pain relief using thoracic epidural analgesia: outstanding success and disappointing failures. Anaesthesia. 2001 Jan;56(1):75-81. doi: 10.1046/j.1365-2044.2001.01763-7.x. PMID 11167441
- [Background] Dolin SJ, Cashman JN, Bland JM. Effectiveness of acute postoperative pain management: I. Evidence from published data. Br J Anaesth. 2002 Sep;89(3):409-23. PMID 12402719
- [Background] Tzimas P, Prout J, Papadopoulos G, Mallett SV. Epidural anaesthesia and analgesia for liver resection. Anaesthesia. 2013 Jun;68(6):628-35. doi: 10.1111/anae.12191. PMID 23662750
- [Background] Koea JB, Young Y, Gunn K. Fast track liver resection: the effect of a comprehensive care package and analgesia with single dose intrathecal morphine with gabapentin or continuous epidural analgesia. HPB Surg. 2009;2009:271986. doi: 10.1155/2009/271986. Epub 2009 Dec 15. PMID 20029637
- [Background] Yong BH, Tsui SL, Leung CC, Lo CM, Liu CL, Fan ST, Young K. Management of postoperative analgesia in living liver donors. Transplant Proc. 2000 Nov;32(7):2110. doi: 10.1016/s0041-1345(00)01592-x. No abstract available. PMID 11120091
- [Background] Koruk M, Onuk MD, Akcay F, Savas MC. Serum thrombopoietin levels in patients with chronic hepatitis and liver cirrhosis, and its relationship with circulating thrombocyte counts. Hepatogastroenterology. 2002 Nov-Dec;49(48):1645-8. PMID 12397754
- [Background] Lin MC, Wu CC, Ho WL, Yeh DC, Liu TJ, P'eng FK. Concomitant splenectomy for hypersplenic thrombocytopenia in hepatic resection for hepatocellular carcinoma. Hepatogastroenterology. 1999 Mar-Apr;46(26):630-4. PMID 10370587
- [Background] Ho AM, Lee A, Karmakar MK, Samy W, Lai PB, Ho OA, Cho A. Hemostatic parameters after hepatectomy for cancer. Hepatogastroenterology. 2007 Jul-Aug;54(77):1494-8. PMID 17708283
- [Background] De Pietri L, Siniscalchi A, Reggiani A, Masetti M, Begliomini B, Gazzi M, Gerunda GE, Pasetto A. The use of intrathecal morphine for postoperative pain relief after liver resection: a comparison with epidural analgesia. Anesth Analg. 2006 Apr;102(4):1157-63. doi: 10.1213/01.ane.0000198567.85040.ce. PMID 16551916
- [Background] Suc B, Panis Y, Belghiti J, Fekete F. 'Natural history' of hepatectomy. Br J Surg. 1992 Jan;79(1):39-42. doi: 10.1002/bjs.1800790113. PMID 1346582
- [Background] Borromeo CJ, Stix MS, Lally A, Pomfret EA. Epidural catheter and increased prothrombin time after right lobe hepatectomy for living donor transplantation. Anesth Analg. 2000 Nov;91(5):1139-41. doi: 10.1097/00000539-200011000-00018. PMID 11049898
- [Background] Oguro A, Taniguchi H, Daidoh T, Itoh A, Tsukuda N, Takahashi T. Factors relating to coagulation, fibrinolysis and hepatic damage after liver resection. HPB Surg. 1993 Aug;7(1):43-9. doi: 10.1155/1993/91843. PMID 8260434
- [Background] Takita K, Uchida Y, Hase T, Kamiyama T, Morimoto Y. Co-existing liver disease increases the risk of postoperative thrombocytopenia in patients undergoing hepatic resection: implications for the risk of epidural hematoma associated with the removal of an epidural catheter. J Anesth. 2014 Aug;28(4):554-8. doi: 10.1007/s00540-013-1776-4. Epub 2013 Dec 29. PMID 24375285
- [Background] Komatsu T, Kino A, Inoue M, Sowa T, Takahashi K, Fujinaga T. Paravertebral block for video-assisted thoracoscopic surgery: analgesic effectiveness and role in fast-track surgery. Int J Surg. 2014;12(9):936-9. doi: 10.1016/j.ijsu.2014.07.272. Epub 2014 Aug 1. PMID 25091399
- [Background] Komatsu T, Sowa T, Takahashi K, Fujinaga T. Paravertebral block as a promising analgesic modality for managing post-thoracotomy pain. Ann Thorac Cardiovasc Surg. 2014;20(2):113-6. doi: 10.5761/atcs.oa.12.01999. Epub 2013 Feb 28. PMID 23445804
- [Background] Karmakar MK, Booker PD, Franks R. Bilateral continuous paravertebral block used for postoperative analgesia in an infant having bilateral thoracotomy. Paediatr Anaesth. 1997;7(6):469-71. doi: 10.1046/j.1460-9592.1997.d01-118.x. PMID 9365974
- [Background] Wassef MR, Randazzo T, Ward W. The paravertebral nerve root block for inguinal herniorrhaphy--a comparison with the field block approach. Reg Anesth Pain Med. 1998 Sep-Oct;23(5):451-6. doi: 10.1016/s1098-7339(98)90026-8. PMID 9773696
- [Background] Weltz CR, Klein SM, Arbo JE, Greengrass RA. Paravertebral block anesthesia for inguinal hernia repair. World J Surg. 2003 Apr;27(4):425-9. doi: 10.1007/s00268-002-6661-5. PMID 12658486
- [Background] Fahy AS, Jakub JW, Dy BM, Eldin NS, Harmsen S, Sviggum H, Boughey JC. Paravertebral blocks in patients undergoing mastectomy with or without immediate reconstruction provides improved pain control and decreased postoperative nausea and vomiting. Ann Surg Oncol. 2014 Oct;21(10):3284-9. doi: 10.1245/s10434-014-3923-z. Epub 2014 Jul 18. PMID 25034821
- [Background] Klein SM, Bergh A, Steele SM, Georgiade GS, Greengrass RA. Thoracic paravertebral block for breast surgery. Anesth Analg. 2000 Jun;90(6):1402-5. doi: 10.1097/00000539-200006000-00026. PMID 10825328
- [Background] Canto M, Sanchez MJ, Casas MA, Bataller ML. Bilateral paravertebral blockade for conventional cardiac surgery. Anaesthesia. 2003 Apr;58(4):365-70. doi: 10.1046/j.1365-2044.2003.03082_2.x. PMID 12688271
- [Background] Sato N, Sugiura T, Takahashi K, Kato G, Kamada T, Mori Y, Kobayashi Y. [Analgesia with paravertebral block for postoperative pain after thoracic or thoracoabdominal aortic aneurysm repair]. Masui. 2014 Jun;63(6):640-3. Japanese. PMID 24979853
- [Background] Richardson J, Vowden P, Sabanathan S. Bilateral paravertebral analgesia for major abdominal vascular surgery: a preliminary report. Anaesthesia. 1995 Nov;50(11):995-8. doi: 10.1111/j.1365-2044.1995.tb05939.x. PMID 8678263
- [Background] Piccioni F, Fumagalli L, Garbagnati F, Di Tolla G, Mazzaferro V, Langer M. Thoracic paravertebral anesthesia for percutaneous radiofrequency ablation of hepatic tumors. J Clin Anesth. 2014 Jun;26(4):271-5. doi: 10.1016/j.jclinane.2013.11.019. Epub 2014 May 20. PMID 24856797
- [Background] Moussa AA. Opioid saving strategy: bilateral single-site thoracic paravertebral block in right lobe donor hepatectomy. Middle East J Anaesthesiol. 2008 Feb;19(4):789-801. PMID 18630766
- [Background] Cheema SP, Ilsley D, Richardson J, Sabanathan S. A thermographic study of paravertebral analgesia. Anaesthesia. 1995 Feb;50(2):118-21. doi: 10.1111/j.1365-2044.1995.tb15092.x. PMID 7710020
- [Background] Richardson J, Lonnqvist PA, Naja Z. Bilateral thoracic paravertebral block: potential and practice. Br J Anaesth. 2011 Feb;106(2):164-71. doi: 10.1093/bja/aeq378. PMID 21233114
- [Background] Naja Z, Lonnqvist PA. Somatic paravertebral nerve blockade. Incidence of failed block and complications. Anaesthesia. 2001 Dec;56(12):1184-8. doi: 10.1046/j.1365-2044.2001.02084-2.x. PMID 11736777
- [Background] Karmakar MK. Thoracic paravertebral block. Anesthesiology. 2001 Sep;95(3):771-80. doi: 10.1097/00000542-200109000-00033. No abstract available. PMID 11575553
- [Background] Richardson J, Sabanathan S, Jones J, Shah RD, Cheema S, Mearns AJ. A prospective, randomized comparison of preoperative and continuous balanced epidural or paravertebral bupivacaine on post-thoracotomy pain, pulmonary function and stress responses. Br J Anaesth. 1999 Sep;83(3):387-92. doi: 10.1093/bja/83.3.387. PMID 10655907
- [Background] Raveglia F, Rizzi A, Leporati A, Di Mauro P, Cioffi U, Baisi A. Analgesia in patients undergoing thoracotomy: epidural versus paravertebral technique. A randomized, double-blind, prospective study. J Thorac Cardiovasc Surg. 2014 Jan;147(1):469-73. doi: 10.1016/j.jtcvs.2013.09.024. Epub 2013 Nov 1. PMID 24183908
- [Background] Richardson J, Sabanathan S, Shah R. Post-thoracotomy spirometric lung function: the effect of analgesia. A review. J Cardiovasc Surg (Torino). 1999 Jun;40(3):445-56. PMID 10412938
- [Background] Davies RG, Myles PS, Graham JM. A comparison of the analgesic efficacy and side-effects of paravertebral vs epidural blockade for thoracotomy--a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2006 Apr;96(4):418-26. doi: 10.1093/bja/ael020. Epub 2006 Feb 13. PMID 16476698
- [Background] Ding X, Jin S, Niu X, Ren H, Fu S, Li Q. A comparison of the analgesia efficacy and side effects of paravertebral compared with epidural blockade for thoracotomy: an updated meta-analysis. PLoS One. 2014 May 5;9(5):e96233. doi: 10.1371/journal.pone.0096233. eCollection 2014. PMID 24797238
- [Background] Jones B, Jarvis P, Lewis JA, Ebbutt AF. Trials to assess equivalence: the importance of rigorous methods. BMJ. 1996 Jul 6;313(7048):36-9. doi: 10.1136/bmj.313.7048.36. PMID 8664772
- [Background] Piaggio G, Elbourne DR, Altman DG, Pocock SJ, Evans SJ; CONSORT Group. Reporting of noninferiority and equivalence randomized trials: an extension of the CONSORT statement. JAMA. 2006 Mar 8;295(10):1152-60. doi: 10.1001/jama.295.10.1152. PMID 16522836
- [Background] Brittain E, Lin D. A comparison of intent-to-treat and per-protocol results in antibiotic non-inferiority trials. Stat Med. 2005 Jan 15;24(1):1-10. doi: 10.1002/sim.1934. PMID 15532089
- [Background] Grider JS, Mullet TW, Saha SP, Harned ME, Sloan PA. A randomized, double-blind trial comparing continuous thoracic epidural bupivacaine with and without opioid in contrast to a continuous paravertebral infusion of bupivacaine for post-thoracotomy pain. J Cardiothorac Vasc Anesth. 2012 Feb;26(1):83-9. doi: 10.1053/j.jvca.2011.09.003. Epub 2011 Nov 17. PMID 22100213
- [Background] Richardson J, Lonnqvist PA. Thoracic paravertebral block. Br J Anaesth. 1998 Aug;81(2):230-8. doi: 10.1093/bja/81.2.230. No abstract available. PMID 9813528